CLINICAL TRIAL: NCT05563337
Title: Renal Denervation in Hypertensive Women Planning to Become Pregnant
Brief Title: Women Hypertensive and Young-Renal Denervation
Acronym: WHY-RDN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHUBX 2020/56; 2021-A02309-32 (Other: ID RCB)
Record Dates: First submitted 2022-08-24; First posted 2022-10-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-08

CONDITIONS: Arterial Hypertension
Keywords: Renal denervation; Pregnancy; Arterial hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Physician who will perform the renal arteriography and renal denervation in case of randomization in the "renal denervation group" will be different from the cardiologist who will follow the patient throughout the study in order to keep the double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denervation treatment (Experimental)
  Interventions: Procedure: Arteriography and renal denervation
- Control (Sham Comparator)
  Interventions: Procedure: Arteriography without renal denervation

INTERVENTIONS:
Procedure: Arteriography and renal denervation — Diagnostic renal Arteriography - Randomization - Renal denervation
  Arms: Denervation treatment
Procedure: Arteriography without renal denervation — Diagnostic renal Arteriography - Randomization
  Arms: Control

SUMMARY:
Renal denervation is a new method to lower blood pressure (BP) in hypertensive patients by reducing the impact of sympathetic nervous system. Its efficacy has been demonstrated in resistant hypertension and in lowering BP in essential hypertension as compared to a sham procedure in untreated hypertensive patients. This procedure is safe without any serious adverse events. However its effects during pregnancy are unknown.

Normal pregnancy is associated with an increase of sympathetic activity at rest and upon cardiovascular reflexes stimulation which returns to baseline after delivery. These changes maintain optimal utero placental blood flow. But excessive stimulation of sympathetic activity may play a role in preeclampsia. Drugs that may affect the sympathetic nervous system are considered as safe in pregnant women.

So there are reasonable evidence that renal denervation performed before pregnancy should not have deleterious effects for the fetus. The efficiency of renal denervation being greater in young patient and in women, a greater proportion of BP normalization can be expected in this population of young women .

DETAILED DESCRIPTION:
Investigators will include women with essential hypertension, treated or untreated, who are planning a short term pregnancy (D0). If high blood pressure is confirmed by ABPM after one month without treatment (D30), investigators will proceed to the arteriography during which they will be randomized in the renal denervation group or in the control one.

After the randomization, BP monitoring by Home BP measurement will be performed every month and send to the investigator. Then the patient will benefit from a new ABPM two months after the intervention (D100), and she may stop contraception and may become pregnant. BP will be monitored during pregnancy by home BP and by a new ABPM at the beginning of the 6th month of pregnancy as well as one, one month after delivery. From the D100, the patient will be able to start an antihypertensive treatment at any time depending on HBPM or ABPM.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years and ≤ 40 years
* Free, informed, written consent signed by the participant and the investigating physician (no later than the day of inclusion and before any examination required by the research)
* Not pregnant but planning to be pregnant in the near future (<2 years)
* Patient using effective contraception, preferably micro-progestational, during the screening phase and the two-month post-procedure follow-up
* Essential hypertension confirmed and documented by a previous complete search
* Hypertension treated by 0-2 antihypertensive treatment(s) in a stable manner for at least 4 weeks and whose clinical BP measured in the sitting position during consultation is ≤ 180/110mmHg at the selection visit (D0),
* Person able to understand and agree to follow all study procedures
* Person who is affiliated or beneficiary of a social security plan

Non-Inclusion Criteria:

* Males of any age
* Females whose age is <18 years or >40
* Orthostatic hypotension
* Hypertension from secondary causes (other than sleep apnea)
* Documented contraindication or proven severe allergy to iodinated contrast
* Contraindication to use anticoagulants
* Renal insufficiency with GFR estimated at < 60ml/min/1.73m²
* Antihypertensive treatment with more than two active ingredients
* Type 1 diabetes or uncontrolled type II diabetes (plasma HbA1c level ≥ 9%)
* History of chronic inflammatory bowel disease such as Crohn's disease or ulcerative colitis
* Brachial circumference > 40 cm
* Any history of a cerebrovascular event (stroke, transient ischemic attack)
* Any history of a serious cardiovascular event (myocardial infarction, acute heart failure requiring hospitalization, coronary artery bypass surgery)
* Proven and confirmed episodes of stable or unstable angina in the 12 months preceding consent
* Proven history of persistent or permanent atrial fibrillation
* Presence of an active implantable medical device (e.g. neuromodulator/spinal modulator, baroreflex stimulator, ...)
* Oxygen therapy or permanent ventilation other than CPAP for sleep apnea
* Primary pulmonary hypertension
* Limited life expectancy (< 1 year)
* Unresolved history of drug or alcohol abuse
* Not have sufficient ability to understand or follow instructions
* In the investigator's opinion she is unlikely to be willing or able to comply with the requirements of the study protocol or participation in the study will involve confounding factors in the analysis of the data
* Participation in another trial of an investigational drug or device (participation in a non-interventional study is tolerated)
* Pregnant or nursing mother
* Person unable to give informed consent
* Person deprived of liberty by judicial or administrative decision
* Adults under legal protection

Exclusion Criteria:

* BP ≤ 135/85 mmHg and ≥ 160/100 mmHg (ABPM) after 4 weeks washout/run-in period.
* Renal arterial anatomy not compatible with renal denervation confirmed by a good quality renal artery angioscan performed within one year prior to consent.
* Patient without at least one artery on each side that can be treated with 2 or more ablations,
* Renal artery anatomy:

  * Main renal artery diameter < 3.0 mm and > 8 mm
  * Main renal artery length < 20 mm
  * A single functioning kidney (low differentiation or small kidney)
  * Kidney tumors presence
  * Renal arterial aneurysm presence
  * Pre-existing renal stent or history of renal artery angioplasty
  * Pre-existing aortic stent or history of aortic aneurysm
  * Prior renal denervation procedure
  * Fibromuscular dysplasia of the renal arteries
  * Presence of renal artery stenosis of any origin ≥ 30%
  * Presence of iliac/femoral artery calcification or stenosis precluding insertion of the Paradise Catheter
  * Infection within 7 days of the procedure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-05-18 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Normalization of 24h blood pressure | at Day 100
  Percentage of patients cured of their hypertension (cure defined as 24h BP<130/80 mmHg at Day 100 without treatment)

SECONDARY OUTCOMES:
Number of adverse events | between Day 0 and 70 months
  Number of adverse events following denervation compared to the control procedure between Day 0 and 1 month after end of pregnancy ( 70 months maximum)
Number of potential pregnancy complications | between Day 0 and 70 months
  Number of potential pregnancy complications between Day 0 and 1 month after end of pregnancy ( 70 months maximum)
Comparison of 24-hour ABPM variations | between Day 30 and 70 months
  Comparison of 24-hour ABPM variations between Day 30 and 1 month after end of pregnancy ( 70 months maximum)
Comparison of Home BP variations | between Day 30 and 70 months
  Comparison of Home BP variations between Day 30 and 1 month after end of pregnancy ( 70 months maximum)
Number of antihypertensive treatments used | at Day 100

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GOSSE, MD, Study Director — University Hospital, Bordeaux
Locations (6):
- France (6):
  - CHU de Bordeaux - Hôpital Saint-André, Bordeaux
  - CHU Grenoble-Alpes, Grenoble
  - CHRU de LILLE - Hôpital Cardiologique, Lille
  - CHU de Nantes - Hôpital Laennec, Nantes
  - APHP - Hôpital Européen Georges-Pompidou, Paris
  - CHU de TOULOUSE - Hôpital Rangueil, Toulouse

REFERENCES:
- [Derived] Gosse P, Sentilhes L, Boulestreau R, Doublet J, Gaudissard J, Azizi M, Cremer A; WHY-RDN investigators. Endovascular ultrasound renal denervation to lower blood pressure in young hypertensive women planning pregnancy: study protocol for a multicentre randomised, blinded and sham controlled proof of concept study. BMJ Open. 2023 Sep 29;13(9):e071164. doi: 10.1136/bmjopen-2022-071164. PMID 37775290